CLINICAL TRIAL: NCT02945345
Title: Evaluation of Clinical Responsiveness Using the Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI)
Brief Title: Clinical Responsiveness of Dermatomyositis Using Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI)
Acronym: CDASI
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Victoria Werth, MD and Principal Investigator, University of Pennsylvania
Other Study IDs: 808230
Record Dates: First submitted 2012-02-09; First posted 2016-10-26 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Dermatomyositis
MeSH Terms: conditions — Dermatomyositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, skin tissue biopsies
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
The Evaluation of Clinical Responsiveness Using the Cutaneous Dermatomyositis Disease Area and Severity Index (CDASI), established in 2008, is a one-site database study conducted at the University of Pennsylvania. The database has yielded valuable information and clinical insights into the pathophysiology, disease processes, including psychological responses, treatments and quality of life associated with dermatomyositis. The CDASI database incorporates the Cutaneous Dermatomyositis Disease Area and Severity Index), a validated outcome measure of disease responsiveness in patients, and other assessment tools, surveys and patient information to help validate the clinical course and quality of life of patients with dermatomyositis.

The CDASI database has led to publication of comparison studies of CDASI and other clinical instruments and the effect of dermatomyositis on Quality of Life (QoL).

The CDASI database is an ongoing resource that enables clinicians to evaluate the evolving clinical changes, treatment modalities and patient response to a challenging disease. Data will be analysed over a 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Gender/Age: Males or females above 18 years old
* Diagnosis: Cutaneous Dermatomyositis
* Subjects able to give informed consent

Exclusion Criteria:

* Subjects without cutaneous DM
* Penn employees
* Penn students
* Cognitively impaired persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have been diagnosed with dermatomyositis.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2008-06 (Actual); Primary Completion 2030-01-02 (Estimated); Study Completion 2030-01-02 (Estimated)

PRIMARY OUTCOMES:
Cutaneous Dermatomyositis Disease Area and Severity Index | through study completion, an average of 1 year
  Disease severity tool

SECONDARY OUTCOMES:
Skin quality of life tool | through study completion, an average of 1 year
  Quality of life tool

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States